CLINICAL TRIAL: NCT06964282
Title: Comparison Between Iliopsoas Block (IPB) and Pericapsular Nerve Group (PENG) Block on Postoperative Analgesia and Functional Recovery After Total Hip Arthroplasty Surgery: a Double-blinded Randomized Clinical Trial
Brief Title: Iliopsoas (IPB) and Pericapsular Nerve Group (PENG) Blocks Comparison on Analgesia and Recovery After Total Hip Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, Michele Carella, Clinical Professor, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-172
Record Dates: First submitted 2025-04-30; First posted 2025-05-09 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Total Hip Arthroplasty (THA); Postoperative Pain Management; Peripheral Nerve Blocks; PENG Block; Iliopsoas Nerve Block

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind, controlled equivalence trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient, the surgeon, and the postoperative data collector will be blinded to the allocation. Only the anesthesiologist performing the block (who is not involved in patient follow-up or data collection) will know the specific technique and dosage used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group PENG (Active Comparator): Patients will receive a pericapsular nerve group block with 14 ml of ropivacaine 3.75 mg/ml, administered 30 minutes prior to spinal anesthesia.
  Interventions: Procedure: PENG Block
- IPB Group (Active Comparator): Patients will receive an iliopsoas plane block with 7 ml of ropivacaine 7.5 mg/ml, administered 30 minutes prior to spinal anesthesia.
  Interventions: Procedure: Iliopsoas nerve block

INTERVENTIONS:
Procedure: PENG Block — Also performed under ultrasound guidance with an 80 mm B-Braun X360 needle and a 3-5 MHz curved probe. The femoral nerve, femoral artery, iliopsoas muscle, and pubic ramus are identified. The needle is inserted in-plane, and 14 ml of ropivacaine 3.75 mg/ml is injected between the psoas tendon and pubic ramus.
  Arms: Group PENG
Procedure: Iliopsoas nerve block — Performed under ultrasound guidance with a curvilinear probe (5-2 MHz). The transducer is positioned transversely below the anterior superior iliac spine (ASIS), then pivoted medially. After identifying the femoral head and acetabular rim, a 22G 80 mm needle is inserted in-plane to reach the iliopsoas plane, lateral to the iliopsoas tendon. 7 ml of ropivacaine 7.5 mg/ml is then injected.
  Arms: IPB Group

SUMMARY:
Background:

In recent years, regional anesthesia has become more popular because it can reduce pain and the need for strong pain medications like morphine. For hip surgery, the PENG block is already known to be effective. A newer method, called the iliopsoas plane block (IPB), is very similar and has also shown good results in hip arthroscopy. However, these two techniques have never been directly compared in patients undergoing hip replacement surgery using the posterior approach.

Goal:

This study aims to see if the IPB is just as effective as the PENG block for controlling pain and helping patients recover well after hip replacement surgery.

Method:

118 adult patients scheduled for hip replacement under spinal anesthesia will be randomly assigned to receive either: IPB: 7 ml of Ropivacaine 7.5 mg/ml PENG: 14 ml of Ropivacaine 3.75 mg/ml Both injections are given under ultrasound guidance 30 minutes before spinal anesthesia. Neither the patient, the surgeon, nor the data collector will know which technique was used.

Post-Surgery Care:

All patients will receive standard pain relief, including:

Paracetamol every 6 hours Etoricoxib once a day Morphine via a patient-controlled pump for 48 hours

Main Outcome Measured:

The primary goal is to compare pain during movement 6 hours after surgery, using a pain scale from 0 (no pain) to 10 (worst pain). The study will consider the two blocks equivalent if the difference in average pain scores is less than 1 point.

Other Outcomes:

Total morphine used in 48 hours Pain scores at rest and during movement at various time points Walking ability (2- and 6-minute walk tests, and timed-up-and-go test) Quality of recovery (using the QoR-15 questionnaire) Side effects of morphine Patient satisfaction Length of hospital stay

Safety:

Both techniques are safe and already used in clinical practice. Ultrasound guidance minimizes risks like nerve injury, bleeding, or infection.

Conclusion:

If the IPB is shown to be as effective as the PENG block, both can be considered reliable options for pain control and early recovery after hip replacement surgery.

DETAILED DESCRIPTION:
This study investigates the comparative effectiveness of two regional anesthesia techniques-the Pericapsular Nerve Group (PENG) block and the Iliopsoas Plane Block (IPB)-in patients undergoing total hip arthroplasty (THA) via the posterior surgical approach. While both blocks have shown promise in managing postoperative pain and minimizing opioid use, direct comparisons between them in this surgical context are lacking.

The PENG block, which targets the articular branches of the femoral, obturator, and accessory obturator nerves, has become increasingly used in anterior and lateral hip surgeries. The IPB, though more recently introduced, involves injection in a similar anatomical region and has shown good analgesic results in patients undergoing hip arthroscopy. Given their overlapping targets, these two blocks may offer comparable clinical benefits; however, this has not been validated in THA performed through a posterior approach.

To address this gap, the current randomized, double-blind equivalence trial will compare the two techniques using standardized ultrasound-guided procedures and uniform dosing of ropivacaine adjusted for volume and concentration. All patients will receive the same spinal anesthetic and postoperative analgesia regimen, minimizing confounding factors.

The primary objective is to determine whether IPB provides pain control equivalent to the PENG block during early postoperative mobilization. By assessing patient-reported pain scores, along with recovery quality and opioid use, the study aims to generate evidence that may inform anesthesia planning in joint replacement surgeries and support the integration of newer regional techniques into enhanced recovery protocols.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (age >18 years) ASA physical status classification I-III Scheduled for elective posterior approach total hip arthroplasty (THA) under spinal anesthesia

Exclusion Criteria:

Pregnancy (confirmed by beta-HCG test if applicable) Known peripheral neuropathy or major neurological disease Chronic pain syndromes or long-term opioid use (>20 mg oral morphine equivalents/day) Severe hepatic or renal insufficiency Allergy to local anesthetics Major coagulopathies Vulnerable patients (e.g., minors, legally protected individuals)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Dynamic Pain 6h postoperative | 6 hours after surgery
  Dynamic pain score (during mobilization) at 6 hours postoperatively, measured on a 0-10 numeric rating scale (NRS). Equivalence is defined as a mean difference of less than 1 point on the NRS.

SECONDARY OUTCOMES:
Total Morphine Consumption | First postoperative 48 hours
  Total morphine consumption at 48 hours on Patient Controlled Intravenous Analgesia device.
NRS Dynamic pain | First postoperative 48 hours
  NRS Dynamic pain score (at tight flexion) at 6 hours postoperatively, measured on a 0-10 numeric rating scale (NRS) and at 8 am, 1 pm, 6pm at postoperative day 1 and day 2. No pain: 0; Maximum pain: 10.
NRS Rest pain | First postoperative 48 hours
  NRS Rest pain score (no mobilization) at 6 hours postoperatively, measured on a 0-10 numeric rating scale (NRS) and at 8 am, 1 pm, 6pm at postoperative day 1 and day 2. No pain: 0; Maximum pain: 10.
2MWT | First postoperative 48 hours
  Distance walked in meters during 2-minute at postoperative day 1 and day 2
6MWT | First postoperative 48 hours
  Distance walked in meters during 6-minutes test at postoperative day 1 and day 2
TUG | First postoperative 48 hours
  Timed Up and Go (TUG) test results at postoperative day 1 and day 2
QoR-15 | First postoperative 48 hours
  Patient recovery scores using the 15-item Quality of Recovery (QoR-15) questionnaire on postoperative days 1 and 2. Minimum: 0; Maximum: 150.
IPO | 48 hours after surgery
  Patient satisfaction using the International Pain Outcomes (IPO) questionnaire at discharge. Each question is a 0 to 10 NRS scale with 0 minimum value and 10 maximum value.
Morphine-related complications | First postoperative 48 hours
  Incidence of opioid-related side effects (nausea, vomiting, constipation, urinary retention, pruritus, dizziness, hypotension)
LOS | 48 hours after surgery
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Michele Carella, MD, PhD, ESRA-DRA, Principal Investigator — Liège University Hospital
Locations (1):
- Liege University Hospital, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No
Patient data will be anonymized and collected via the REDCap platform, compliant with current data protection regulations. Only the principal investigator and authorized study personnel will have access. Data will be stored securely for 10 years.